CLINICAL TRIAL: NCT07377747
Title: Prospective Study Evaluating the Treatment Outcomes for Localised Recurrent, Resectable Retroperitoneal Liposarcoma
Acronym: ReLaPSe
Status: Recruiting | Type: Observational
Sponsor: Australia and New Zealand Sarcoma Association (Other)
Responsible Party: Sponsor
Other Study IDs: X23-0316
Record Dates: First submitted 2026-01-04; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Retroperitoneal Liposarcoma
Keywords: Sarcoma; liposarcoma; retroperitoneal
MeSH Terms: conditions — Retroperitoneal liposarcoma; Sarcoma; Liposarcoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery with preoperative radiotherapy: This includes patient who have had any chemotherapy.
- Surgery without preoperative radiotherapy: This includes patients who had surgery alone, surgery with postoperative radiotherapy and/or any chemotherapy.

SUMMARY:
The aim of the study is to collect prospective data on the treatment outcomes in patients with first localized, resectable recurrent retroperitoneal well-differentiated and/or dedifferentiated liposarcoma undergoing curative intent treatment. Patients enrolled in this study will form a validation cohort of the TARPSWG recurrent RPS nomogram. The treatment decision (surgery alone, or preoperative RT +/- chemotherapy followed by surgery) is per the institutional multidisciplinary team recommendation.

DETAILED DESCRIPTION:
This study is collecting participant data prospectively from hospital medical records. Participant details regarding diagnosis, treatments, outcomes, complications and survival status will be captured after patients are enrolled into the study and at specific time points though out the study. Participants will also be asked to complete quality of life questionnaires called the EORTC QLQ-C30 and the OLO-STO22 at 4 or 5 different time points which will take 15-20 minutes to complete. The overall duration of observation is from time of enrolment for 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Adult age ≥ 18 presenting with first recurrent well-differentiated and/or dedifferentiated liposarcoma of retroperitoneal space or pelvis after previous macroscopically complete resection (R0/R1 resection)
2. No distant metastasis on cross-sectional imaging of chest/abdomen/pelvis (CT and/or MRI) within 1 month to confirm the absence of metastatic disease
3. Previous histologically proven well-differentiated or dedifferentiated liposarcoma histology only
4. Sarcoma not originating from bone or abdominal or gynecological viscera
5. Tumor confirmed to be resectable with likely R0/R1 resection, and all disease must be deemed to be treatable by RT (joint decision by surgeon and radiation oncologist at a sarcoma multidisciplinary team meeting)
6. WHO performance status 0-2
7. American Society of Anaesthesiologist (ASA) score 1-3
8. No prior RT for the retroperitoneal liposarcoma
9. Prior systemic therapy is allowed
10. No concurrent active malignancy (except for low risk skin malignancy, low risk prostate carcinoma, low risk breast carcinoma including in situ disease)
11. Women of childbearing potential must have a negative pregnancy test within 3 weeks prior to the first day of study treatment
12. Patient deemed able to comply with study requirements according to investigator evaluation
13. Signed, IRB-approved written informed consent

Exclusion Criteria:

1. Unresectable disease or likely R2 resection as assessed by the multidisciplinary sarcoma team
2. Extent of recurrence where preoperative RT to all visible disease is not deemed to be feasible
3. Contradiction for RT such as history of bowel obstruction or mesenteric ischemia or severe chronic inflammatory bowel disease
4. Myxoid liposarcoma histology
5. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with localized, resectable recurrent retroperitoneal liposarcoma attending and having treatment at the study site.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Abdominopelvic recurrence-free survival (ARFS). . | Up to 5 years.
  Defined as the time from the date of treatment start (either surgery, chemo or RT) for 1st recurrent LPS to the date of radiological abdominopelvic relapse or death whichever occurred first. Liver metastases will be regarded as distant metastatic events. rather than abdominopelvic relapse

SECONDARY OUTCOMES:
Overall survival | Up to 5 years.
  Overall survival will be measured from the date of treatment start to the date of death, whatever the cause. Alive patients will be censored during the study and at each follow-up visit (usually every 3-6 months) for up to 5 years. Causes of death will be recorded.
Cumulative incidence of 2nd local recurrence (in a competing risk framework) | Up to 5 years.
Cumulative incidence of distant metastases (in a competing risk framework). | Up to 5 years.
Cumulative incidence of in-field relapse for those who had preoperative radiotherapy (in a competing risk framework) | Up to 5 years.
Pathological response using the EORTC-STBSG criteria. | At surgical resection.
  Obtained by using the standardised pathological evaluation score for assessing tumour response as recorded in the patient's medical records.
Radiology response to preoperative RT. | Within 4 weeks of surgery.
  The tumor response will be assessed using RECIST 1.1 and Choi criteria by comparison of baseline cross-sectional imaging (CT-scan or MRI) and preoperative imaging within 4 weeks of surgery (same modality). Response criteria are based on a set of measurable lesions identified at baseline as target lesions and followed at the preoperative imaging performed within 2 weeks of surgery.
Local disease progression during preoperative radiotherapy. | During preoperative radiotherapy (for those patients that have preoperative radiotherapy)
  Local disease progression during preoperative radiotherapy rendering disease no longer operable
Distant disease progression during preoperative RT. | During preoperative radiotherapy (for those patients that have preoperative radiotherapy).
Toxicity of preoperative radiotherapy | From the start of preoperative radiotherapy up to one week prior to surgery
Surgical complication | Up to 60 days post surgery
Health related quality of life using the EORTC QLQ-C30 and the EORTC QLQ-STO22 assessment scales. | At registration, during the last week of RT treatment (preoperative RT patients only), within 2 weeks prior to surgery (for the preoperative RT patients), at 3 months and 12 months after surgery.
  The QLQ-C30 (core questionnaire) and the QLQ-STO22 (gastric cancer-specific module) are used together. Scores range from 0-100 with higher scores meaning better quality of life.
Unplanned R2 resection | At surgery
Stratified analysis of use of chemotherapy | Up to 5 years.
Validation of the recurrent RPS nomogram and the dynamic primary RPS nomogram | Up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hong, Principal Investigator — Chris O'Brien Lifehouse
Locations (9):
- United States (3):
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - OSU James Hospital, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- UZ Leuven, Leuven, Flemish Brabant, Belgium
- A.C.Camargo Cancer Center - Fundacao Antonio Prudente, Liberdade, São Paulo, Brazil
- The Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands